CLINICAL TRIAL: NCT03795597
Title: Phase I/II Study Utilizing High Dose Busulfan and Melphalan With Escalating Carfilzomib as Conditioning in Autologous Peripheral Blood Stem Cell Transplantation for Patients With Multiple Myeloma
Brief Title: Busulfan, Melphalan, Escalating Carfilzomib Conditioning Auto Stem Cell Transplantation for Multiple Myeloma (MM)
Acronym: BuMelCarAuto
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Patrick Stiff, Principal Investigator, Loyola University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 209274
Record Dates: First submitted 2018-10-17; First posted 2019-01-08 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Autologous; Stem Cell Transplantation; Bone Marrow Transplant; Carfilzomib
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Busulfan; Melphalan

STUDY DESIGN:
Intervention Model Description: Busulfan IV over 3 hours every 24 hours for a total of 4 doses from D-6 to D-3. First two daily infusions will be given at a fixed dose of 3.2 mg/kg over 3 hours from D-6 to D-5. The 3rd and 4th daily doses will be adjusted to an AUC of approximately 5,000 mMol-min per dose.
  Melphalan 140 mg/ m2 IV over 15-30 minutes for one dose on day -3.
  Carfilzomib administration will follow a Phase I dose escalation design.
  Each cohort will start with a goal of accruing three patients to determine the dose limiting toxicities.
  Once the Maximum Tolerated Dose is established an expansion cohort will be treated to include a total of 10 additional patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Carfilzomib IV at dose: 20 mg/m2 (Experimental): The participants will receive Carfilzomib IV at dose: 20 mg/m2 on days -9 and -8 over 30 minutes. The participant will receive Busulfan IV over 3 hours every 24 hours for a total of 4 doses from Day -6 to Day -3 and Melphalan IV over 15-30 minutes for one dose on day -3.The participants will receive stem cell infusion on Day 0 and Granulocyte-Colony stimulating factor (G-CSF) given daily until engraftment occurs.
  Interventions: Drug: Carfilzomib; Drug: Busulfan IV; Drug: Melphalan IV
- Carfilzomib IV at dose: 27 mg/m2 (Experimental): The participants will receive Carfilzomib IV at dose: 27 mg/m2 on days -9 and -8 over 30 minutes. The participant will receive Busulfan IV over 3 hours every 24 hours for a total of 4 doses from Day -6 to Day -3 and Melphalan IV over 15-30 minutes for one dose on day -3.The participants will receive stem cell infusion on Day 0 and G-CSF given daily until engraftment occurs.
  Interventions: Drug: Carfilzomib; Drug: Busulfan IV; Drug: Melphalan IV
- Carfilzomib IV at dose: 36 mg/m2 (Experimental): The participants will receive Carfilzomib IV at dose: 36 mg/m2 on days -9 and -8 over 30 minutes. The participant will receive Busulfan IV over 3 hours every 24 hours for a total of 4 doses from Day -6 to Day -3 and Melphalan IV over 15-30 minutes for one dose on day -3.The participants will receive stem cell infusion on Day 0 and G-CSF given daily until engraftment occurs.
  Interventions: Drug: Carfilzomib; Drug: Busulfan IV; Drug: Melphalan IV
- Carfilzomib IV at dose: 45 mg/m2 (Experimental): The participants will receive Carfilzomib IV at dose: 45 mg/m2 on days -9 and -8 over 30 minutes. The participant will receive Busulfan IV over 3 hours every 24 hours for a total of 4 doses from Day -6 to Day -3 and Melphalan IV over 15-30 minutes for one dose on day -3.The participants will receive stem cell infusion on Day 0 and G-CSF given daily until engraftment occurs.
  Interventions: Drug: Carfilzomib; Drug: Busulfan IV; Drug: Melphalan IV
- Carfilzomib IV at dose: 56 mg/m2 (Experimental): The participants will receive Carfilzomib IV at dose: 56 mg/m2 on days -9 and -8 over 30 minutes. The participant will receive Busulfan IV over 3 hours every 24 hours for a total of 4 doses from Day -6 to Day -3 and Melphalan IV over 15-30 minutes for one dose on day -3.The participants will receive stem cell infusion on Day 0 and G-CSF given daily until engraftment occurs.
  Interventions: Drug: Carfilzomib; Drug: Busulfan IV; Drug: Melphalan IV

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib is an anti-cancer drug acting as a selective proteasome inhibitor that is used to treat Multiple Myeloma.
  Other Names: Kyprolis
Drug: Busulfan IV — Busulfan is an anti-cancer drug acting as a bifunctional alkylating agent that is used to treat Multiple Myeloma.
  Other Names: Busulfex
Drug: Melphalan IV — Melphalan is an anti-cancer drug acting as alkylating agent that is used to treat Multiple Myeloma.
  Other Names: Alkeran

SUMMARY:
In this protocol, the investigators hypothesize that the combination of intravenous busulfan and melphalan with carfilzomib will be an effective preparative regimen with acceptable toxicity for participants with multiple myeloma who are candidates for autologous stem cell transplantation. To test this hypothesis, the investigators designed a phase I/II trial combining IV busulfan 130 mg/m2 plus melphalan 140 mg combined with escalating doses of carfilzomib ranging from 20 mg/m2 to 45 mg/m2. These results will be compared with the center's historical controls of participants treated with melphalan, busulfan and bortezomib.

DETAILED DESCRIPTION:
Participants enrolled in this study protocol will receive daily intravenous (IV) infusions of carfilzomib for a total of 4 days (Day-9, -8 and Days -2, -1). The first two daily infusions will be given at a fixed dose of 20 mg/m2 and the final two doses will be escalated from the standard dose of 27 mg/m2 to 56 mg/m2 in a Phase I design, based on toxicity. The busulfan will be administered for 2 days over 3 hours from D-7, -6, at 130 mg/m2 . This dose was found to be safe and equivalent to the standard daily dose of 3.2 mg/kg. The 3rd and 4th daily doses of IV Busulfan will be adjusted in order to yield a systemic plasma drug exposure represented by a daily area under the plasma concentration versus time curve (AUC) of approximately 5,000 millimoles-minute per dose (mM-min). These targeted plasma concentration of IV busulfan will be based on pharmacokinetics studies performed during the first day of IV busulfan. Melphalan will be given at a dose of 140 mg/m2 on Day -3. Each cohort will start with a goal of accruing three patients to determine the dose limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be greater than or equal to 18 years of age.
* Participants must have been diagnosed with multiple myeloma in a first or subsequent remission and have undergone a successful pre-transplant work up and are otherwise eligible for an autotransplant with a busulfan/melphalan preparative regimen at Loyola University Medical Center.
* Participants may receive this preparative regimen if in first or subsequent remission. Participants may enter if they have received a prior autologous stem cell transplant and this therapy produced a remission that lasted greater than 18 months before progression of disease. Participants who have undergone prior allogeneic transplantation are excluded.
* All participants must have responsive disease as defined by a Partial Response or greater to most recent conventional regimen.
* Participants receiving prior carfilzomib will be eligible for inclusion provided they demonstrated responsive disease to this agent and either had a remission that lasted greater than 6 months after its discontinuance, or if in remission after a carfilzomib containing regimen administered to qualify for transplant.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) less than or equal to 2.
* Acceptable heart function test.

Exclusion Criteria:

* Participants must not have below normal kidney function.
* Participants must not have below normal liver function.
* Participants must not have active bacterial, fungal, or viral infection.
* Participants must not have severe lung function.
* Participants must not have Grade 2 or greater peripheral neuropathy.
* Participants must not have uncontrolled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
36 participants evaluated for safety with treatment-related adverse events and grading by using CTCAE v4.0. | 3 years
  To determine the maximal tolerated dose of carfilzomib when added to busulfan and melphalan as a preparative regimen for high dose therapy with autologous hematopoietic transplantation for patients with multiply myeloma.
36 participants evaluated for tolerability with treatment-related adverse events and grading by using CTCAE v4.0. | 3 years
  To determine the maximal tolerated dose of carfilzomib when added to busulfan and melphalan as a preparative regimen for high dose therapy with autologous hematopoietic transplantation for patients with multiply myeloma.

SECONDARY OUTCOMES:
36 participants evaluated for response to treatment by testing blood for multiple myeloma levels. | 100 days
  To evaluate complete, very good partial, partial and stable disease response rate for both clinical and biologic endpoints.
36 participants evaluated for progression by testing blood for multiple myeloma levels. | 3 years
  Progression Free Survival
36 participants evaluated for overall survival by clinical visit or contact by phone. | 3 years
  Overall Survival
36 participants evaluated for absolute neutrophil count by testing white blood cells levels. | 100 days
  Days to neutrophil engraftment: Absolute neutrophil count > 500/microliter
36 participants evaluated for platelet engraftment by testing platelet count in blood cells. | 100 days
  Days to platelet engraftment: platelet count > 20,000/microliter untransfused
36 participants evaluated by oral exam to assess mucositis events and grading levels by using CTCAE v4.0. | 100 days
  Mucositis: CTCAE v 4.0 grade and severity
36 participants evaluated by the liver to assess Veno-occlusive disease and grading levels by using CTCAE v4.0. | 100 days
  Veno-occlusive disease
36 participants evaluated by a physical exam to assess peripheral neuropathy and grading by using CTCAE v4.0. | 3 years
  Peripheral neuropathy greater than or equal to CTCAE V 4.0 Grade 3
36 participants evaluated for response to treatment by testing urine for multiple myeloma levels. | 100 days
  To evaluate complete, very good partial, partial no stable disease response rate for both clinical and biologic endpoints
36 participants evaluated for progression by testing urine for multiple myeloma levels. | 3 years
  Progression Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stiff, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No